CLINICAL TRIAL: NCT00321581
Title: Phase I Trial of CEDIRANIB (AZD2171), an Orally Bioavailable Antiangiogenic Agent, in Children and Adolescents With Refractory or Recurrent Solid Tumors
Brief Title: AZD2171 to Treat Children and Adolescents With Solid Tumors or Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060152; 06-C-0152; NCT00354848 (obsolete NCT alias)
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2012-06-29

CONDITIONS: Refractory or Recurrent Solid Tumors; Acute Myelogenous Leukemia
Keywords: VEGFR2; Tyrosine Kinase Inhibitor; Antiangiogenesis; Solid Tumors; Childhood Cancer; Solid Tumor; Recurrent Solid Tumor; Treatment Resistant Solid Tumor; Acute Myelogenous Leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — cediranib

INTERVENTIONS:
Drug: Cediranib, AZD2171, RECENTIN

SUMMARY:
Background:

* AZD2171 is an experimental drug that may slow the growth of cancers by blocking angiogenesis (formation of new blood vessels).
* Cancer growth is dependent on angiogenesis for nutrition.
* Inhibiting angiogenesis is a new approach to cancer therapy.

Objectives:

* To determine the side effects of AZD2171 in children and adolescents with cancer.
* To determine the highest dose of AZD2171 that can safely be given to children and adolescents with cancer.
* To study how the body handles AZD2171.
* To determine the effects of AZD2171 on various factors related to angiogenesis.
* To determine if AZD2171 can inhibit cancer growth in children and adolescents.

Eligibility:

-Children and adolescents 2-18 years of age with treatment-resistant solid tumor cancers or acute myelogenous leukemia.

Design:

* About 40 patients may be included in the study.
* AZD2171 is given by mouth in treatment cycles of once a day for 28 days. Treatment may continue unless the cancer worsens or unacceptable side effects develop.
* Patients have periodic physical examinations, blood and urine tests and imaging tests (CT, X-rays, MRI) to evaluate disease throughout the course of treatment. Additional blood tests are done to study how the body handles AZD2171, to look for proteins that stimulate angiogenesis, to determine if certain blood vessel cells are affected by AZD2171, and for other research purposes.
* Biopsy tissue (when available) is examined for the receptor for new blood vessel formation.

DETAILED DESCRIPTION:
Background:

* Cediranib is a potent orally bioavailable inhibitor of VEGFR1, VEGFR2, VEGFR3 tyrosine kinase activity, but also inhibits c-kit and PDGFR-Beta in vitro.
* Phase I trials of Cediranib are ongoing in adults and the drug is well tolerated at doses up to 45 mg/d. The toxicity profile includes hypertension, hypoglycemia, elevated LFTs, fatigue, dysphonia, diarrhea, nausea and vomiting.

Objectives:

* To determine the maximum tolerated dose (MTD) and dose-limiting toxicities of orally administered Cediranib on a daily for 28 consecutive days schedule in children and adolescents with refractory childhood solid tumors.
* To define the toxicity spectrum of oral Cediranib in children and adolescents.
* To assess the pharmacokinetics and pharmacodynamics of oral Cediranib in children and adolescents.
* Assess growth plate volume in the right knee using non-contrast MRI scans prior to and during administration of cediranib.

Eligibility:

-Children and adolescents (greater than 2 yrs and less than 19 years of age) with histologically confirmed relapsed or refractory extracranial solid tumors that are measurable or evaluable.

Design:

* Cediranib will be administered orally, daily. Treatment cycles are 28 days with no break in treatment between cycles. The starting dose level is 12 mg/m(2)/d with escalations to 17, 25, 35, and 50 mg/ m(2)/d, due to dose limiting toxicity in the initial 2 subjects enrolled at 12 mg/m(2)/d the protocol was amended to restart dose escalation at 8 mg/m(2)/d.
* Detailed pharmacokinetic and pharmacodynamic studies will be performed during the first 28 day treatment cycle.
* The trial follows a standard phase I design with 3 to 6 patients per dose level and standard definitions of MTD and DLT. Up to 28 patients will be entered on this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

AGE: Patients must be greater than 2 years and less than 19 years of age.

DIAGNOSIS: Solid Tumors (dose escalation component of the trial): Histologically confirmed extracranial malignant solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing's sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, and germ cell tumors.

DISEASE STATUS: Patients with solid tumors must have measurable or evaluable disease.

- Patients must be able to swallow tablets intact.

PRIOR THERAPY: The patient's cancer must have relapsed after or failed to respond to frontline standard therapy and no other standard curative treatment options are available. Standard therapy may include surgery, radiation therapy, chemotherapy, or any combination of these modalities.

Patients must have had their last fraction of radiation therapy:

* at least 4 months prior to study entry for large ports (greater than 50% pelvis, TBI, or craniospinal) for solid tumor patients.
* at least 4 weeks prior to study entry for other radiation in solid tumor patients or for any type of radiation in leukemia patients.

Patients must have had their last dose of:

Cytotoxic chemotherapy:

-Patients with solid tumors, the last dose of cytotoxic therapy must be at least 21 days prior to study entry.

Biological therapy that was administered for the treatment of cancer at least 7 days prior to study entry.

Immunotherapy (antibody) at least 30 days prior to study entry.

Any investigational cancer therapy at least 30 days prior to study entry.

Patients who have received an allogeneic BM or SC transplant must be at least 3 months post-transplant; and patients who have received an autologous BM or SC transplant must be at least 2-months post-transplant.

Patients must have recovered from the acute toxic effects of prior therapy before entry onto this trial.

Patients should be off colony stimulating factors such as filgrastim (G-CSF), sargramostim (GM-CSF), and IL-11 (with the exception of erythropoietin) for at least 72 hours prior to study entry. Patients receiving PEG-filgrastim (Neulasta ) must be at least 7 days from the last dose.

CONCOMITANT MEDICATIONS:

* Patients requiring systemic full dose anticoagulation with systemic thrombolytics, heparin, coumadin, low molecular weight heparin, or other anticoagulants for therapy of active thrombosis within the prior 3 months are excluded.
* Patients receiving prophylactic anticoagulation for thrombosis are eligible if they meet criteria for adequate hemostatic function (PT and PTT less than or equal to 1.5 x ULN) and the thrombotic episode occurred greater than 3 months prior to enrollment. Use of anticoagulants or thrombolytics for care and maintenance of central venous catheters (e.g., intralumenal TPA) is acceptable.
* Patients on thyroid replacement (levothyroxine, synthroid ) must be on a stable dose for at least 1 month.
* Patient receiving a medication that has a known risk of QTc prolongation with in the last 2 weeks are excluded.
* Patient receiving corticosteroids must be on a stable or tapering dose for 14 days prior to study enrollment.

PERFORMANCE STATUS: Patients greater than 10 years old must have a Karnofsky performance level greater than 50, and children less than or equal to 10 years old must have a Lansky performance level greater than 50.

HEMATOLOGICAL FUNCTION:

-Patients with solid tumors must have adequate bone marrow function, defined as a peripheral absolute neutrophil count of greater than or equal to 1,500/microL, and a platelet count greater than or equal to 100,000/microL (transfusion independent).

Coagulation: Patients must have adequate hemostatic function defined as PT and PTT less than or equal to 1.5 x ULN. It is recommended that PT and PTT be drawn by peripheral venipuncture rather than from an indwelling central venous catheter.

CARDIAC: Patients must have:

* QTc (Bazett's Correction) less than or equal to 480 msec on ECG.
* Normal Left Ventricular Diastolic Function: Echocardiogram with ejection fraction greater than or equal to 55 percent or shortening fraction greater than or equal to 27 percent.

HEPATIC FUNCTION: Patients must have adequate liver function, defined as bilirubin less than or equal to 1.5 x ULN, SGPT (ALT) less than or equal to 2.5 x ULN.

RENAL FUNCTION:

* Proteinuria less than or equal to 1 + on dipstick when urine specific gravity is less than or equal to 1.015 or 24 hr urine total protein is less than or equal to 500 grams/24hr.
* Patients must have an age-adjusted normal serum creatinine (See Table Below) OR a creatinine clearance is greater than or equal to 60 mL/min/1.73 m(2).

  2 to less than 6 years of age equals a maximum serum creatinine of 0.8 mg/dl.

  6 to less than 10 years of age equals a maximum serum creatinine of 1 mg/dl.

  10 to less than 13 years of age equals a maximum serum creatinine of 1.2 mg/dl.

  13 years to less than 16 years of age equals a maximum serum creatinine of 1.5 mg/dl (male) and 1.4 mg/dl (female).

Greater than or equal to 16 years of age equals a maximum serum creatine of 1.7 mg/dl (male) and 1.4 mg/dl (female).

INFORMED CONSENT: All patients or their legal guardians (if the patient is less than 18 years old) must sign a document of informed consent (Pediatric Oncology Branch, NCI screening protocol for NIH patients) prior to performing studies to determine patient eligibility. After confirmation of patient eligibility all patients or their legal guardians must voluntarily sign the IRB approved protocol specific informed consent to document their understanding of the investigational nature and the risks of this study before any protocol related studies are performed (other than the studies which were performed to determine patient eligibility).

DURABLE POWER OF ATTORNEY (DPA): Patients who are 18 years of age will be offered the opportunity to assign a DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

BIRTH CONTROL: Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are receiving protocol therapy and for 2 weeks after the last dose of Cediranib.

EXCLUSION CRITERIA:

Patients with primary brain tumors.

Patients with a history of congenitally prolonged QTc, or history of arrhythmia (multifocal premature ventricular contractions, bigeminy,trigeminy, ventricular tachycardia, uncontrolled atrial fibrillation, left bundle block) that is symptomatic or requires treatment (except for controlled atrial fibrillation).

* Patients receiving medication for treatment of hypertension or patients with a diastolic blood pressure 5mmHg greater than the 95% for gender and age on 3 measurements using an appropriate size cuff are excluded.
* Patients who have had major surgery within the past 3 months. Patients having minor surgery (e.g., central line placement) within the past 2 weeks.
* Patients with history of arterial or venous thrombosis within the prior 3 months.
* Patients requiring systemic full dose anticoagulation with systemic thrombolytics, heparin, coumadin, or low molecular weight heparin or other anticoagulants for therapy of active thrombosis within the prior 3 months.
* Patients experiencing significant hemorrhage (hemoptysis, melena, or hematemesis) within the past 2 weeks.
* Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal, gastrointestinal or other organ dysfunction, which in the judgment of the principal investigator, protocol chairperson or associate investigator would compromise the patient's ability to tolerate the investigational agent or are likely to interfere with the study procedures or endpoints.
* Patients with active GVHD are excluded.
* Pregnant or breastfeeding females are excluded because Cediranib may be harmful to the developing fetus or nursing child.
* Patients currently receiving other investigational agents.
* Patients previously known to be Hepatitis B, Hepatitis C, or HIV infected because of the unknown interaction of Cediranib with antiviral therapy.
* Patients or first degree relatives of persons that are involved in the planning and conduct of this trial are excluded.
* Patients who have previously received Cediranib.
* Patients who are allergic to Cediranib or its excipients (mannitol, sodium starch glycollate and magnesium stearate).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05-01; Study Completion 2011-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Childrens Hospital, Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Folkman J. What is the evidence that tumors are angiogenesis dependent? J Natl Cancer Inst. 1990 Jan 3;82(1):4-6. doi: 10.1093/jnci/82.1.4. No abstract available. PMID 1688381
- [Background] Arap W, Pasqualini R, Ruoslahti E. Cancer treatment by targeted drug delivery to tumor vasculature in a mouse model. Science. 1998 Jan 16;279(5349):377-80. doi: 10.1126/science.279.5349.377. PMID 9430587
- [Background] Konerding MA, Malkusch W, Klapthor B, van Ackern C, Fait E, Hill SA, Parkins C, Chaplin DJ, Presta M, Denekamp J. Evidence for characteristic vascular patterns in solid tumours: quantitative studies using corrosion casts. Br J Cancer. 1999 May;80(5-6):724-32. doi: 10.1038/sj.bjc.6690416. PMID 10360650
- [Derived] Fox E, Aplenc R, Bagatell R, Chuk MK, Dombi E, Goodspeed W, Goodwin A, Kromplewski M, Jayaprakash N, Marotti M, Brown KH, Wenrich B, Adamson PC, Widemann BC, Balis FM. A phase 1 trial and pharmacokinetic study of cediranib, an orally bioavailable pan-vascular endothelial growth factor receptor inhibitor, in children and adolescents with refractory solid tumors. J Clin Oncol. 2010 Dec 10;28(35):5174-81. doi: 10.1200/JCO.2010.30.9674. Epub 2010 Nov 8. PMID 21060028